CLINICAL TRIAL: NCT06082505
Title: A Community Based Program to Increase Breast and Cervical Cancer Screening and HPV Vaccination to Reduce the Impact of Breast and Cervical Cancer Among Latinas.
Brief Title: Salud en Mis Manos - Breast and Cervical Cancer Prevention and Early Detection - Expansion 1
Acronym: SEMM1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, Lara Savas, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HSC-SPH-16-0159; PP160047 (Other Grant/Funding Number: Cancer Prevention and Research Institute of Texas)
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-10

CONDITIONS: Cervical Cancer; Breast Cancer
Keywords: Cervical cancer prevention; Breast cancer detection; HPV vaccination
MeSH Terms: conditions — Uterine Cervical Neoplasms; Breast Neoplasms | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Person Delivered Breast and Cervical Cancer Behavioral Intervention (Experimental): Community health worker deliver behavioral education and referrals to low-cost services. Deliver in person to participants in community and clinic settings. Participants are followed up by health coach navigators to address barriers and connect to safety-net clinics.
  Interventions: Behavioral: Education; Behavioral: Navigation to clinic
- Telephone Delivered Breast and Cervical Cancer Behavioral Intervention (Experimental): Community health worker deliver behavioral education and referrals to low-cost services. Participants are followed up by health coach navigators to address barriers and connect to safety-net clinics.
  Interventions: Behavioral: Education; Behavioral: Navigation to clinic

INTERVENTIONS:
Behavioral: Education — Education will be delivered in person in a group education setting or individually by phone. Group education will include 1 hour breast and cervical cancer prevention education session delivered with support of electronic presentations. For phone education, trained project staff or Community Health Workers (CHWs) will deliver telephone-based education as an alternative to group education session for women who missed scheduled session twice (education materials would be printed and mailed).
Behavioral: Navigation to clinic — Continue telephone based navigation tailored to participants' barriers using the Cancer Prevention Plan of Action to support, problem solve, assist, and provide reminders to increase utilization of clinic services.

SUMMARY:
The purpose is to evaluate implementation of a community-based prevention project aimed at increasing early detection and prevention of breast and cervical cancer through education and navigation and to increase breast and cervical cancer screening and Human Papillomavirus (HPV) vaccination in underserved Latinas.

DETAILED DESCRIPTION:
This is an evaluation of the Salud en Mis Manos community health worker-delivered breast and cervical cancer screening promotion program. The investigators evaluate the effect of the program on increasing participant breast and cervical cancer screening and HPV vaccination, using a one-group pre-post study design (March 2017 - May 2019). The investigators also describe the implementation of the program during a longer time period (November 2016 - May 2019).

ELIGIBILITY:
Inclusion Criteria:

* Self identifies as Hispanic or Latina
* Lives in Texas
* Breast cancer screening group: have not had a mammogram in the past 2 years, and are 40 years of age and older
* Cervical cancer screening group: have not had a Pap test in the past 3 years and are 21 years of age and older
* HPV vaccination group: are women 21-26 years of age, and have not initiated the HPV vaccine series
* Age limit for breast cancer screening group: 40 years and older
* Age limit for cervical cancer screening group (Pap test): 21 years and older
* Age limit for HPV vaccination group: 21-26 years

Exclusion Criteria:

* Current pregnancy
* Current or prior cancer diagnosis

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8262 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Number of women 40 years and older who complete mammogram screening | Between baseline and end of study (about 9 months)
  Among women 40 years and older that have not had a mammogram in the past two years, enrolled in the program and completed baseline and follow-up surveys.
Number of women 21-65 years old who complete Pap test screening | Between baseline and end of study (about 9 months)
  Among women 21 - 65 years old that have not had a Pap test in the past three years, enrolled in the program and completed baseline and follow-up surveys.
Number of women 21-26 years old who initiate their HPV vaccination series. | between baseline and end of study (about 9 months)
  Among women 21-26 years old that have not yet initiated their HPV vaccination series, enrolled in the program and completed baseline and follow-up surveys.

SECONDARY OUTCOMES:
Number of participants who received the second dose of HPV vaccine | between baseline and end of study (about 9 months)
  Among women that have not had their second HPV vaccination dose, enrolled in the program and completed baseline and follow-up surveys.
Number of participants who received the third dose of HPV vaccine | between baseline and end of study (about 9 months)
  Among women that have not had their third HPV vaccination dose, enrolled in the program and completed baseline and follow-up surveys.
Number of participants who received a clinical breast exam | between baseline and end of study (about 9 months)
  Among women that have not had a mammogram in the past two years, enrolled in the program and completed baseline and follow-up surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Savas, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No